CLINICAL TRIAL: NCT04092322
Title: Validation of Physical Activity Scale for the Elderly (PASE) in Stroke Patients: Relationship Between PASE and Physical Activity Measured by Portable Accelerometer
Brief Title: Validation of Physical Activity Scale for the Elderly (PASE) in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.205
Record Dates: First submitted 2019-09-15; First posted 2019-09-17 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-09

CONDITIONS: Stroke
Keywords: stroke; physical activity; accelerometer; physical activity scale for elderly
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with subacute chronic stroke: Patients with subacute chronic stroke between the ages of 40-80
  Interventions: Device: Actical accelerometers (Philips Respironics); Other: PASE

INTERVENTIONS:
Device: Actical accelerometers (Philips Respironics) — patients with stroke will be evaluated by using PASE scale and accelerometer results (accelerometer will be held from Monday to Friday
Other: PASE — Physical Activity Scale for Elderly

SUMMARY:
The Physical Activity Scale for the Elderly (PASE) is a self-report questionnaire on exercise, home, and work-related physical activities performed during the last week. PASE has shown to be reliable and valid in different populations of people between 65 and 100 years of age and after stroke. However, its validation on stroke was based on another self report questionnaire that assess physical activity called ''Senior Fitness Test''. Since accelerometers are more objective methods to assess PA, to the best of our knowledge, self-report physical activity questionnaires should be validated based on accelerometer derived physical activity data. The aim of this study is to validate PASE in patients with stroke based on accelerometer data.

DETAILED DESCRIPTION:
The Physical Activity Scale for the Elderly (PASE) is a self-report questionnaire on exercise, home, and work-related physical activities performed during the last week. PASE has shown to be reliable and valid in different populations of people between 65 and 100 years of age and after stroke. However, its validation on stroke was based on another self report questionnaire that assess physical activity (PA) called ''Senior Fitness Test''. There are four methods to measure physical activity: 1. Self-Report Questionnaires 2.Self-Report Activity Diaries/Logs 3.Direct Observation 4. Devices (Accelerometers, pedometers, arm band, Heart-Rate Monitors). Accelerometers can measure PA accurately and have ability capture large amounts of data. Accelerometers measure acceleration (activity counts:AC) in real time and detect movement in up to three orthogonal planes (anteroposterior, mediolateral, and vertical) These counts are then translated into a metric of interest, which can be biological (e.g. energy expenditure) or PA patterns (e.g. stationary). There are pros and cons of measurement methods of physical activity. Strengths of accelerometers include minute-by-minute on-line monitoring, capturing intensity level. Accumulated AC provide an accurate estimate of the duration and intensity of body movement at the waist and were summed across the whole day to assess total PA volume. However, accelerometers are expensive and require technical expertise, specialized hardware, software, and individual programming. Self-report PA measurement methods are able to measure large numbers of participants at low cost. Since accelerometers are more objective methods to assess PA, to the best of our knowledge, self-report physical activity questionnaires should be validated based on accelerometer derived physical activity data. The aim of this study is to validate PASE in patients with stroke based on accelerometer data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with first ever, unilateral stroke
2. Patients with stroke who can walk independently or with an assistive device
3. Being at between the ages of 40-80

Exclusion Criteria:

1. Illiteracy
2. Having severely impaired mental function and being unable to complete questionnaires
3. Presence of neglect, demantia, apraxia
4. Having uncontrolled hypertension, cardiopulmonary disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke between the ages of 40-80 who can walk independently or with an assistive device
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
PASE | Day 0
  Physical Activity Score for Elderly

SECONDARY OUTCOMES:
ACtotal | Day 0
  Total activity count obtained from accelerometer
EE total | Day 0
  Total energy expenditure obtained from accelerometer
AC moderate | Day 0
  activity counts derived from accelerometer during moderate physical activity
EE moderate | Day 0
  energy expenditure obtained from accelerometer during moderate physical activity
AC light | Day 0
  activity counts derived from accelerometer during light physical activity
EE light | Day 0
  energy expenditure obtained from accelerometer during light physical activity
AC vigorous | Day 0
  activity counts derived from accelerometer during vigorous physical activity
EE vigorous | Day 0
  energy expenditure obtained from accelerometer during vigorous physical activity
AC sedentary | Day 0
  activity counts derived from accelerometer during sedentary physical activity
EE sedentary | Day 0
  energy expenditure obtained from accelerometer during sedentary physical activity
step count | Day 0
  total step count obtained from accelerometer
Stroke Impact Scale total score | Day 0
  Stroke Impact Scale is a stroke specific quality of life scale. The current version of the SIS (SIS version 3.0) is a 59-item patient-reported outcome measure, covering 8 domains: strength (4 items), hand function (5 items), mobility (9 items), activities of daily living (10 items), memory (7 items), communication (7 items), emotion (9 items), and handicap (8 items). Domains are scored on a metric of 0 to 100, with higher scores indicating better self-reported health. Four of the scales of the SIS can be combined into a composite physical domain (strength, hand function, physical and instrumental activities of daily living, and mobility), with scores also presented on a 0 to 100 metric.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Karadag Saygi, Prof, Study Chair — Marmara University; Esra Giray, MD, Principal Investigator — Marmara University; Nurullah Eren, PT, Principal Investigator — Marmara University School of Health Sciences
Locations (1):
- Esra Giray, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marianne Lindahl, Lotte Hansen, Anders Pedersen, Thomas Truelsen & Gudrun Boysen (2008) Self-reported physical activity after ischemic stroke correlates with physical capacity, Advances in Physiotherapy, 10:4, 188-194, DOI: 10.1080/14038190802490025
- [Result] Hills AP, Mokhtar N, Byrne NM. Assessment of physical activity and energy expenditure: an overview of objective measures. Front Nutr. 2014 Jun 16;1:5. doi: 10.3389/fnut.2014.00005. eCollection 2014. PMID 25988109
- [Result] Persson CU, Hansson PO, Lappas G, Danielsson A. Physical Activity Levels and Their Associations With Postural Control in the First Year After Stroke. Phys Ther. 2016 Sep;96(9):1389-96. doi: 10.2522/ptj.20150367. Epub 2016 Mar 24. PMID 27013578
- [Result] Sylvia LG, Bernstein EE, Hubbard JL, Keating L, Anderson EJ. Practical guide to measuring physical activity. J Acad Nutr Diet. 2014 Feb;114(2):199-208. doi: 10.1016/j.jand.2013.09.018. Epub 2013 Nov 28. No abstract available. PMID 24290836